CLINICAL TRIAL: NCT01446133
Title: Combination of Lenalidomide and Rituximab in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL-SLL) as Initial Treatment or Subsequent Therapy
Brief Title: Combination of Lenalidomide and Rituximab in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL-SLL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0509; NCI-2012-01119 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Leukemia; Lymphoma
Keywords: Leukemia; Lymphoma; Chronic Lymphocytic Leukemia; CLL; Small Lymphocytic Lymphoma; SLL; Initial Treatment; Subsequent Therapy; Rituximab; Rituxan; Lenalidomide; CC-5013; Revlimid
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Untreated 65 + (Experimental): Patients with untreated SLL/CLL with indications for treatment that are age 65 or older.
  Rituximab (375 mg/m2) will be given intravenously on Day 1, Day 8, Day 15 and Day 22 and then continued once every 4 weeks during cycles 3-12 (+ 7 days). Rituximab will not be given in Cycle 2. Lenalidomide will be started on Day 9 of cycle 1 at the dose of 10 mg/day and will be continued daily. Treatment duration will be 12 cycles and it will be possible to continue beyond 12 cycles if there is a significant benefit such as an ongoing Partial Response or Complete Response.
  Interventions: Drug: Rituximab; Drug: Lenalidomide
- Prior Treatment Any Age (Experimental): Patients of any age with previously treated CLL/SLL and recurrent disease.
  Rituximab (375 mg/m2) will be given intravenously on Day 1, Day 8, Day 15 and Day 22 and then continued once every 4 weeks during cycles 3-12 (+ 7 days). Rituximab will not be given in Cycle 2. Lenalidomide will be started on Day 9 of cycle 1 at the dose of 10 mg/day and will be continued daily. Treatment duration will be 12 cycles and it will be possible to continue beyond 12 cycles if there is a significant benefit such as an ongoing Partial Response or Complete Response.
  Interventions: Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 by vein on Day 1, Day 8, Day 15 and Day 22 and then continued once every 4 weeks during cycles 3-12 (+ 7 days). Rituximab will not be given in Cycle 2.
  Other Names: Rituxan
Drug: Lenalidomide — 10 mg/day by mouth daily beginning on Day 9 of cycle 1.
  Other Names: CC-5013; Revlimid

SUMMARY:
The goal of this clinical research study is to learn if the combination of lenalidomide and rituximab can help to control CLL. The safety of this drug combination will also be studied.

Lenalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. This may decrease the growth of cancer cells.

Rituximab is designed to attach to cancer cells and damage them, which may cause the cells to die.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will begin taking the study drugs in 28-day cycles. One time a week during Cycle 1, you will receive rituximab by vein. During Cycle 2, you will not receive rituximab. During Cycles 3-12, you will receive rituximab on Day 1 of Cycles 3-12. Your first dose of rituximab will be given over 6-8 hours. If you tolerate your first dose well, you may receive the next doses over 2-4 hours. If the doctor thinks it is needed, the next doses may given over a longer time.

Starting on Day 9 of Cycle 1, you will begin taking lenalidomide by mouth 1 time a day.

The dose and schedule of lenalidomide may change depending on the side effects you may have. You should swallow lenalidomide capsules whole with a glass (8 ounces) water at the same time each day. Do not break, chew, or open the capsules. If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss a dose, it should NOT be made up on another day.

During Cycle 1 only, you will take allopurinol by mouth 1 time a day on Days 1-14 to lower the risk of side effects.

Study Visits:

One (1) time a week during the first 5 weeks, blood (about 1 tablespoon) will be drawn for routine tests.

After the first 5 weeks, blood (about 1 tablespoon) will be drawn for routine tests every 2 weeks until the doctor thinks your dose of lenalidomide can stay the same. After that, blood (about 1 tablespoon) will be drawn every 4 weeks for the rest of the study for routine tests.

At the end of Cycles 3, 6, and 12, you will have a bone marrow biopsy and aspiration to check the status of the disease.

If you stay on study past 12 cycles, once every 6 cycles (Cycles 18, 24, 30, and so on), you will have a bone marrow biopsy and aspiration to check the status of the disease.

Blood (about 1 tablespoon) will be drawn more often if the dose of lenalidomide needs to be changed or if you have intolerable side effects.

Pregnancy Testing:

If you are able to become pregnant, you will have a urine or blood (less than 1 teaspoon) pregnancy test 10-14 days and 24 hours before the first dose of lenalidomide, even if you have not had a menstrual period due to treatment of the disease or had only 1 menstrual period in the past 24 months.

If you have regular or no menstrual cycles, you will then have a urine or blood (less than 1 teaspoon) pregnancy test every week for the first 4 weeks, then every 4 weeks while taking lenalidomide, again as soon as you stop taking lenalidomide, and then 28 days after you have stopped taking lenalidomide.

If you have irregular menstrual cycles, you will have a urine or blood (less than 1 teaspoon) pregnancy test every week for the first 4 weeks, then every 2 weeks while taking lenalidomide, again as soon as you stop taking lenalidomide, and then at 14 days and 28 days after you have stopped taking lenalidomide.

Length of Treatment:

You may receive rituximab for up to 12 cycles. You may continue taking lenalidomide for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed your last study drug dose (if you are male) or your last follow-up pregnancy test (if you are female).

This is an investigational study. Lenalidomide and rituximab are FDA approved and commercially available. Lenalidomide is approved for the treatment of multiple myeloma and some myelodysplastic syndromes. Rituximab is approved for the treatment of CLL. The combination of these drugs to treat CLL is investigational.

Up to 120 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/-18 at the time of signing of informed consent.Understand and voluntarily sign informed consent.
2. Patients with chronic lymphocytic leukemia and untreated disease with indication for treatment that are not candidates or unwilling to receive chemoimmunotherapy, or patients of any age with previously treated CLL/SLL or recurrent disease. Patients with recurrent disease are eligible if they have received prior treatment with purine analog based chemotherapy or chemoimmunotherapy or bendamustine.
3. ECOG/WHO performance status of 0-2.
4. Adequate renal function indicated by serum creatinine less or equal to 2mg/dL
5. Adequate hepatic function indicated as total bilirubin less or equal to 2mg/dL and ALT less or equal to 2 times the upper limit of normal.
6. Disease free of prior malignancies for 3 years with exception of current basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast. Patients with malignancies with indolent behavior such as prostate cancer treated with radiation or surgery can be enrolled in this study as long as they have a reasonable expectation to have been cured with the treatment modality received.
7. All study participants must be registered into the mandatory RevAssist program and be willing and able to comply with the program requirements.
8. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mlU/mL within 10-14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1. Prescriptions must be filled within 7 days and must either commit to continued abstinence from heterosexual intercourse or use two acceptable methods of birth control, one highly effective method and one additional effective method at the same time at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

Exclusion Criteria:

1. Known sensitivity to lenalidomide or other thalidomide derivatives or rituximab.
2. Documented prolymphocytic leukemia (prolymphocytes more than 55% in the peripheral blood).
3. Known positivity for HIV or active hepatitis B or C.
4. Pregnant or breast feeding females.
5. History of tuberculosis treated within the last five years or recent exposure to tuberculosis.
6. Any serious medical condition, laboratory abnormality, or psychiatric illness that places the subject at unacceptable risk if he/she were to participate in the study.
7. Patients with a recent history of deep vein thrombosis (DVT) or pulmonary embolus (PE) in the six months prior to enrollment are not eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-12-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 6 months
  Participants evaluated for response by 2008 International Workshop on Chronic Lymphocytic Leukemia [IWCLL] overall response criteria by 6 months of treatment. Bone marrow biopsy and aspiration to check the status of the disease. Responses assessed after 3, 6 and 12 cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, MD,BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Strati P, Takahashi K, Peterson CB, Keating MJ, Thompson PA, Daver NG, Jain N, Burger JA, Estrov Z, O'Brien SM, Kantarjian HM, Wierda WG, Futreal PA, Ferrajoli A. Efficacy and predictors of response of lenalidomide and rituximab in patients with treatment-naive and relapsed CLL. Blood Adv. 2019 May 14;3(9):1533-1539. doi: 10.1182/bloodadvances.2019031336. PMID 31076409
- [Derived] Takahashi K, Hu B, Wang F, Yan Y, Kim E, Vitale C, Patel KP, Strati P, Gumbs C, Little L, Tippen S, Song X, Zhang J, Jain N, Thompson P, Garcia-Manero G, Kantarjian H, Estrov Z, Do KA, Keating M, Burger JA, Wierda WG, Futreal PA, Ferrajoli A. Clinical implications of cancer gene mutations in patients with chronic lymphocytic leukemia treated with lenalidomide. Blood. 2018 Apr 19;131(16):1820-1832. doi: 10.1182/blood-2017-11-817296. Epub 2018 Jan 22. PMID 29358183
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org